CLINICAL TRIAL: NCT01796509
Title: Multicenter Randomised, Controlled Trial of a Intensive Care Follow -up Programme in Improving Long-term Outcomes of ICU Survivors
Brief Title: Study in Intensive Care Follow-up Programme in Improving Long-term Outcomes of ICU Survivors
Acronym: SUIVI-REA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P100147
Record Dates: First submitted 2013-02-13; First posted 2013-02-21 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-02

CONDITIONS: Quality of Life; Post ICU Discharge
Keywords: Quality of life,; Sequela disorders,; Socio-professional impact,; Anxiety, depression,; Post traumatic stress disorder,; ICU acquired paresis.
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multidisciplinary follow-up (Experimental)
  Interventions: Other: Medical, psychological, social
- no follow-up (No Intervention)

INTERVENTIONS:
Other: Medical, psychological, social — After having given his consent, the patient filled auto questionnaire, and then randomized either in follow up arm (i.e. intervention group) or in no follow up arm (i.e. control group). In the follow up arm, medical, psychological and social consultation will be planned within the first seven days after inclusion, and then 3, 6, 12 months. During medical consultation a general examination will be performed, muscle strength, cognitive function, functional disabilities will be assessed with help of MRC, MMS. During psychological consultation, anxiety and depression will be assessed with the help of HAD, IES. The psychologist will also have a free interview. During social consultation personal and professional reinsertion will be assessed.
  Arms: multidisciplinary follow-up

SUMMARY:
Study Hypothesis:

Critical illness is associated with long-term medical and psychological sequelae that can impact the professional and private life. The purpose of the present multicenter randomized controlled trial is to assess whether or not a medical, psychological and social follow-up improves quality of life of critically ill patients at one year after their discharge from intensive care unit (ICU).

Primary Purpose:

Death or severe alteration of quality of life assessed with help of EQ5D questionnaire at one year after ICU discharge.

DETAILED DESCRIPTION:
Critically ill patients who had required at least 3 days of mechanical ventilation and who consented to participate will be randomized at time of ICU discharge in either follow-up or not follow-up arm. The medical, psychological and social follow-up consists of multidisciplinary consultation at time of ICU discharge (i.e. inclusion), at three, six and 12 months afterward. Patients of the "non follow-up group" will be seen only at one year. Medical consultation will be focused on evaluation of pre-existing co-morbidities, detection of new ones and of physical disorders related to critical illness (i.e. ICU-acquired paresis, pain, functional disability, cognitive dysfunction…). Psychological assessment will be focused on detection of anxiety, depression and post-traumatic stress syndrome. Social follow-up will assess the social need of the patient in the professional and private domains. Each assessment will be standardized by using validated or appropriate scores. At the end of each multidisciplinary consultation, a report will be sent to the patient and his general practitioner. When necessary, a consultation with a specialist will be organized. At one year, an observer blinded from randomization will call all the patients to assess their quality of life with help of EQ5D questionnaire. Economical cost of multidisciplinary follow-up will be assessed.

To our knowledge, there is no follow-up studies that have combined a medical, psychological and social cares. For instance, the PracTical study has not evidenced an improvement of quality of life in patients who had beneficiated from nurse consultations at 3 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18
* Living in an area near the hospital
* Hospitalized in the ICU medical surgical hospitals in this study.
* Who required mechanical ventilation more than 3 days
* Having a life expectancy greater than one year (Mc Cabe score >2, absence of metastatic cancer)
* Having a general practitioner identified
* Is affiliated to a social health care
* And who have given their written informed consent

Exclusion Criteria:

* Patients hospitalized in ICU in the previous year
* Patients followed for a preexisting myopathy
* The burn patients, patients with brain injury (Glasgow initial <8) or trauma
* Patients hospitalized for suicide or self-induced poisoning
* Patients with psychiatric disorders
* Patients with ore dementia
* Pregnant women
* Patients who do not speak fluently French
* Patients with guardianship
* Homeless patients
* No having a general practitioner identified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Death or severe alteration of quality of life assessed after ICU discharge | 1 year
  Death or severe alteration of quality of life assessed with help of EQ5D questionnaire at one year after ICU discharge.

SECONDARY OUTCOMES:
Assessment of life quality in Medical domain | 1 year
  ICU-acquired paresis assessed with help of MRC sum score, Functional disabilities assessed with help of Barthel and IADL scales, Cognitive dysfunctions assessed with help of MMS score, Pain, Comorbidities (Hypertension, etc…).
Assessment in psychological domain | 1 year
  Anxiety assessed with help of HAD scale, Depression assessed with help of HAD scale Post-traumatic stress syndrome assessed with help of IES scale.
Assessment in social domain | 1 year
  Social reinsertion with help of RNLI scale.
Assessment in economical cost | 1 year
  Number of hospitalization,number of outpatient consultation and prescription of new treatment will be assessed within 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Sharshar, MD, PHD, Study Director — ICU, Hôpital Raymond Poincaré; Diane Friedman, MD, Principal Investigator — ICU, Hôpital Raymond Poincaré
Locations (1):
- Hôpital Raymond Poincaré, Garches, Île-de-France Region, France

REFERENCES:
- [Derived] Friedman D, Grimaldi L, Cariou A, Aegerter P, Gaudry S, Ben Salah A, Oueslati H, Megarbane B, Meunier-Beillard N, Quenot JP, Schwebel C, Jacob L, Robin Lagandre S, Kalfon P, Sonneville R, Siami S, Mazeraud A, Sharshar T. Impact of a Postintensive Care Unit Multidisciplinary Follow-up on the Quality of Life (SUIVI-REA): Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2022 May 9;11(5):e30496. doi: 10.2196/30496. PMID 35532996